CLINICAL TRIAL: NCT00128960
Title: Prospective Assessment of Functional Status, Psychosocial Adjustment, Health Related Quality of Life and the Symptom Experience in Patients Treated With Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Quality of Life in Patients Who Have Undergone Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 050216; 05-CC-0216
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-04-04

CONDITIONS: Long Term Psychological Affects on HSCT
Keywords: Allogeneic Hematopoietic Stem Cell Transplant; Health Related Quality of Life; Symptom Experience; Fatigue; Functional Status; Natural History
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Participants with different types of diseases and conditions who have undergone an allogeneic (donor) stem cell transplant.

SUMMARY:
This study will evaluate the long-term functional status, psychosocial adjustment and quality of life of patients with different types of diseases and conditions who have had an allogeneic (donor) stem cell transplant. Information from this study may help patients and families know better what they may expect long-term after transplant and will help health care workers improve services to aid in patients' recovery.

People 18 years of age or older who have had an allogeneic stem cell transplant three or more years before the start of this study may be eligible to participate.

Participants complete a series of questionnaires once a year for three years. The questionnaires take about 40 minutes to complete and include information on patient demographics, patients' physical, social, and emotional functioning, spiritual well being, pain, mental health, general health, fatigue, and other areas of health-related quality of life. The questionnaires are completed at home or during normally scheduled follow-up visits to the NIH.

DETAILED DESCRIPTION:
Clinical research in allogeneic hematopoietic stem cell transplantation (HSCT) documents improvements in disease free intervals, disease free survival, and the severity of treatment related toxicities. Those who survive, however, continue to experience side-effects and psychological difficulties for years following allogeneic HSCT. Long term complications occur as delayed effects of the conditioning regimen and the transplant as well as side effects from medications required to maintain the new donor-derived immune system. In addition to various biological complications, long-term effects on the psychological, social, physical, functional and symptoms experience (growth and limitations) have been documented.

Although some knowledge exists to help us understand the experience of various groups of allogeneic HSCT patients, the face of allogeneic transplant has changed considerably over the last five years and limits the application of existing reports. Patients with new types of diseases e.g. solid tumor and those who are older (greater than 55 years) and with more significant debilitation are undergoing allogeneic HSCT. It is important for patients and families to know the effects they can expect following an allogeneic transplant. This lack of clarity of the research limits our ability to focus future intervention studies to begin making a difference for patients at high risk for poor health outcomes following allogeneic HSCT.

Understanding of factors associated with variability in recovery following allogeneic HSCT can increase the likelihood that patients will ultimately return to a normal, productive life. Existing research regarding the recovery of adult survivors of allogeneic HSCT indicates that many patients experience difficulties in a variety of Health Related Quality of Life (HRQL) domains. A critical issue which has remained unexamined concerns the extent to which domains improve, remain static, or perhaps even deteriorates with the passage of time after allogeneic HSCT. Results will be discussed with respect to their implications for both the encouragement of realistic expectations for recovery following allogeneic HSCT as well as the development of interventions.

The long term goal of this study is to characterize longitudinally the functional health, psychosocial adjustment, HRQL and symptom experience associated with long term survival after allogeneic HSCT. This study has two specific aims:

1. To examine the functional status, psychosocial adjustment and HRQL of patients greater than or equal to 3 years following allogeneic HSCT.
2. To examine the symptom experience of patients greater than or equal to 3 years following allogeneic HSCT.

Data will be analyzed using methods of longitudinal analysis, such as the generalized estimating equations, mixed-effects models and growth mixture modeling to evaluate change over time for each outcome variable.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients surviving three years or more from the date of first allogeneic HSCT provided at the Clinical Center, NIH.

Age greater than or equal to 18 years old.

Ability to comprehend the investigational nature of the study and provide informed consent.

Able to read and speak English or Spanish.

Life expectancy of at least 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NIH Clinical Center patients who have undergone allogeneic stem cell transplant.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2005-08-11 (Actual)

PRIMARY OUTCOMES:
Characterize Longitudinally the functional health, psychosocial Adjustment, HRQL and symptom experience associated with LT Survival after allogeneic HSCT. | 3 yrs
  Quality of Life
To examine the symptom experience of patients following allogeneic HSCT | 3 yrs
  Quality of Life

SECONDARY OUTCOMES:
examine functional status, psychosocial adjustment, HRQL, and the symptom experience of patients = 3 years from their transplant as related to late and persistent effects (e.g. complications) of allogeneic HSCT. | 3 years after HSCT
  description of functional status, psychosocial adjustment, HRQL, and the symptom experience

CONTACTS AND LOCATIONS:
Overall Officials: Sandra A Mitchell, C.R.N.P., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bevans MF, Mitchell SA, Barrett JA, Bishop MR, Childs R, Fowler D, Krumlauf M, Prince P, Shelburne N, Wehrlen L, Yang L. Symptom distress predicts long-term health and well-being in allogeneic stem cell transplantation survivors. Biol Blood Marrow Transplant. 2014 Mar;20(3):387-95. doi: 10.1016/j.bbmt.2013.12.001. Epub 2013 Dec 17. PMID 24355521
- [Background] Bevans MF, Mitchell SA, Barrett AJ, Bishop M, Childs R, Fowler D, Krumlauf M, Prince P, Shelburne N, Wehrlen L. Function, adjustment, quality of life and symptoms (FAQS) in allogeneic hematopoietic stem cell transplantation (HSCT) survivors: a study protocol. Health Qual Life Outcomes. 2011 Apr 17;9:24. doi: 10.1186/1477-7525-9-24. PMID 21496339
- [Background] Prince P, Mitchell SA, Wehrlen L, Childs R, Savani B, Yang L, Bevans M. Spiritual Well-Being in Hispanic and Non-Hispanic Survivors of Allogeneic Hematopoietic Stem Cell Transplantation. J Psychosoc Oncol. 2015;33(6):635-54. doi: 10.1080/07347332.2015.1082167. PMID 26315721
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-CC-0216.html